CLINICAL TRIAL: NCT01804049
Title: Metformin and Muscle in Insulin-resistant Older Veterans
Acronym: M&M
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLIN-019-12S
Record Dates: First submitted 2013-02-28; First posted 2013-03-05 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Prediabetes
Keywords: metformin; muscle; insulin resistance; sarcopenia; older adults; impaired fasting glucose
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Sarcopenia | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 60 participants will be randomized to placebo pills.
  Interventions: Drug: placebo
- Metformin (Active Comparator): 60 enrolled participants will be randomized to metformin.
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — Metformin will be given at a dose of 850 mg orally once daily for 1 month with titration up to 850 mg orally twice daily for the remainder of the study.
  Other Names: Glucophage
  Arms: Metformin
Drug: placebo — One placebo capsule by mouth once daily for 1 month followed by one placebo capsule by mouth twice daily for the remainder of the study.
  Arms: Placebo

SUMMARY:
Sarcopenia is the loss of muscle mass, strength and function with aging and is associated with increased disability, falls and fractures. Older adults with diabetes and prediabetes are insulin resistant and have a higher risk of developing sarcopenia. This study examines the use of metformin, an antidiabetic drug, for preventing the development of sarcopenia in older adults with prediabetes.

DETAILED DESCRIPTION:
The proposed study utilizes clinical and translational research approaches to study sarcopenia. Sarcopenia is common in older adults and is associated with decreased strength, increased disability, falls and fractures. There are currently few interventions to prevent or treat sarcopenia and a poor understanding of the mechanisms for sarcopenia. Given the growing number of Veterans over the age of 65, studies to prevent sarcopenia and resulting disability are important for the health, independence and well-being of this population. The investigators' preliminary studies have shown that older adults with diabetes have an accelerated loss in muscle mass and gait speed, except when treated with metformin. Older adults with prediabetes also have a greater decline in muscle mass and higher incidence of disability. Therefore, this study further investigates these findings by addressing the following aims: (1) to determine whether metformin can prevent the loss in muscle mass and physical performance and (2) to examine changes in muscle histologic characteristics associated with metformin treatment in older adults with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will enroll 120 sedentary, weight-stable, ambulatory Veterans aged 65 years and older with prediabetes identified with fasting glucose values 100 mg/dL or greater but under 126 mg/dL with no use of diabetes medications.
* Participants must demonstrate that they are able to ambulate 400 meters without assistance.

Exclusion Criteria:

* Chronic medical conditions affecting muscle mass or function like active non-skin cancer and hypogonadism
* Medications affecting muscle mass or function like glucocorticoids and androgen/antiandrogens
* Contraindications to metformin such as renal dysfunction defined as creatinine >= 1.5 mg/dL for men or >=1.4 mg/dL for women or estimated glomerular filtration rate (eGFR)<60 mL/min; liver dysfunction defined as alanine aminotransferase (ALT)>48 U/L, aspart aminotransferase (AST)>41 U/L or alkaline phosphatase (AlkPhos)>141 U/L; B12 deficiency defined as B12 level <180 pg/dL; congestive heart failure; known hypersensitivity to metformin; excessive alcohol intake (average of 2 or more alcoholic beverages/day over a month)

For the muscle biopsy substudy, additional exclusion criteria include:

* Conditions that include bleeding risk such as the use of warfarin, clopidogrel/ticlopidine, aggrenox, dabigatran or anagrelide; laboratory results showing platelets<150 billion/L or international normalized ratio (INR)>1.2 or activated partial thromboplastin time (aPTT)>36 seconds
* Allergy to lidocaine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Klein, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via advertisement flyers, primary care referral and letters to subjects in the research data warehouse within the Portland VA Healthcare System between May 2014 and August 2015. The first participant was enrolled in the study on May 27,2014 and the last participant was enrolled on August 12, 2015.
Pre-assignment Details: Of the 431 assessed for eligibility, 120 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 43 | 77
Completed | 32 | 45
Not Completed | 11 | 32
Not completed — Adverse Event | 2 | 10
Not completed — Lost to Follow-up | 2 | 1
Not completed — Decreased interest/personal | 4 | 5
Not completed — Other health concerns | 2 | 7
Not completed — Moved out of area | 0 | 7
Not completed — other MD recommended | 1 | 1
Not completed — Enrollment in dual studies | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 43 | 77 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (6.5) | 71.2 (5.1) | 71.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 39 | 76 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 42 | 71 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.527 (4.177) | 29.246 (4.860) | 29.347 (4.610)
Dual-energy X-ray absorptiometry (DEXA) Total Lean Mass (g) [Mean (Standard Deviation); unit: grams] | 58902.9 (7882.7) | 59412.4 (7366.0) | 59227.8 (7526.4)
DEXA Appendicular Lean Mass (g) [Mean (Standard Deviation); unit: grams] | 24676.7 (3913.7) | 24923.5 (3599.3) | 24834.0 (3700.7)
400 Meter Walk Time (seconds) [Mean (Standard Deviation); unit: seconds] | 292.9 (50.2) | 297.3 (48.8) | 295.7 (49.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Lean Mass From Baseline
Description: At baseline, 1, 2, and 3 year follow-up visits, participants will have whole body dual x-ray absorptiometry scans (DXA) with a Hologic QDR 4500W DXA scanner by a certified DXA operator to determine total body lean mass and appendicular lean mass (Kg). The changes in appendicular and total lean mass were calculated by determining the change from baseline to the three year data point. If participants withdrew from the study prior to collection of 3 year data, the final time point available was used.
Time Frame: 3 years
Population: A simple adaptive randomization scheme was developed to balance gender, age and BMI. 120 subjects were randomized to treatment conditions according to 64% to 36% allocation probabilities. Subjects were followed for up to 3 years, with walk time and lean mass measured annually. The study experienced roughly 38% loss-to-follow up at year 3.
Measure: Geometric Mean (Standard Deviation); unit: grams lean mass
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 77
grams lean mass
  Appendicular Lean Mass Decrease from Baseline | 322.8 (1342.3) | 697.6 (2318.8)
  Total Lean Mass Decrease from Baseline | 392.4 (2583.8) | 548.0 (2339.4)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority — Hypothesis: metformin will reduce loss of total lean mass in insulin-resistant older adults over a three year period. It was determined (prior to the initiation of the study) that a sample size of 60 participants per group will have a 73% power to detect a 0.09 m/s difference in gait speed; p = 0.45, t-test, 2 sided — For lean total body mass, t(118)=0.744, p=0.45; T-test calculation for total lean mass: 0.74
Statistical Analysis 2: Comparison: Placebo vs Metformin; Test type: Superiority — Hypothesis: metformin will reduce loss of total appendicular lean mass in insulin-resistant older adults over a three year period. It was determined (prior to the initiation of the study) that a sample size of 60 participants per group will have a 73% power to detect a 0.09 m/s difference in gait speed; p = 0.79, t-test, 2 sided — For lean appendicular body mass, t(118) = 0.264, p=0.79; T-test calculation appendicular lean mass: 0.26

2. Secondary Outcome: Change in Physical Performance - 400 Meter Walk Speed
Description: At baseline, 1, 2, and 3 year follow-up visits, participants will have physical performance assessed using a 400 meter timed walk. We report the 400 meter timed walk speed as the change from baseline in seconds. The change in walk speed from baseline to the three year time point was used for analysis. For participants who withdrew from the study early, the walk speed from the final data point collected was used.
Time Frame: 3 years
Measure: Geometric Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 43 | 77
seconds | -2.82 (51.35) | 0.46 (29.98)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority; p = 0.48, t-test, 2 sided; t(118)=0.703, p=0.48

3. Secondary Outcome: Change in Muscle Characteristics
Description: At baseline and 6 month follow-up visits, 32 subjects will undergo a muscle biopsy of the vastus lateralis muscle 15 cm above the patella using the modified Bergstrom technique under local anesthesia. The muscle biopsy specimens will be used for the histochemical and transcriptome analyses
Time Frame: 6 months
Population: Due to loss of sample and unmatched (time 0 and 6 month) sample availability as well as poor sample integrity, no interpretable histology data is available. No histology data was collected/analyzed from any samples for this Outcome measure.
Groups:
- Placebo: A subgroup of the main study consented to muscle biopsy at time 0 and 6 months of the study. 13 participants were randomized to the placebo biopsy substudy. Placebo was administered as per the main study.
- Metformin: A subgroup of the main study consented to muscle biopsy at time 0 and 6 months of the study. 19 participants were randomized to the metformin biopsy substudy. Metformin was administered as per the main study.
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a three year period.
Description: At each study visit, participants were queried regarding adverse events. In between visits, participants could contact study staff to notify staff of adverse events. Laboratory tests were collected at participant visits and were evaluated for adverse events by study staff.
Groups:
- Placebo: 60 participants were to be randomized to placebo pills.
  placebo: One placebo capsule by mouth once daily for 1 month followed by one placebo capsule by mouth twice daily for the remainder of the study.
  43 participants were allocated to the placebo group.
- Metformin: 60 enrolled participants were to be randomized to metformin.
  metformin: Metformin will be given at a dose of 850 mg orally once daily for 1 month with titration up to 850 mg orally twice daily for the remainder of the study.
  77 participants were allocated to the metformin group.
Arm/Group | Placebo | Metformin
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/77
Serious Adverse Events (participants affected / at risk) | 25/43 | 52/77
Other Adverse Events (participants affected / at risk) | 24/43 | 52/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | Metformin (N=77)
small bowel obstruction (Gastrointestinal disorders) | 1 | 0
pancreatitis (Gastrointestinal disorders) | 0 | 1
stroke/TIA (Nervous system disorders) | 0 | 2
prostatectomy (Surgical and medical procedures) | 1 | 5
abscess (Infections and infestations) | 0 | 1
atrial fibrillation (Cardiac disorders) | 1 | 1
appendicitis (Infections and infestations) | 0 | 1
rectal bleeding (Gastrointestinal disorders) | 0 | 1
syncope (Nervous system disorders) | 0 | 2
acute kidney injury (Renal and urinary disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 1 | 2
chest pain (Cardiac disorders) | 1 | 4
altered mental status (Nervous system disorders) | 1 | 0
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 3
acute cholecystitis (Gastrointestinal disorders) | 1 | 1
elective craniotomy (Surgical and medical procedures) | 0 | 1
transsphenoidal pituitary surgery (Surgical and medical procedures) | 1 | 0
hip replacement (Surgical and medical procedures) | 1 | 0
leukemia (Blood and lymphatic system disorders) | 0 | 1
severe anemia (Blood and lymphatic system disorders) | 0 | 1
large hematoma (Injury, poisoning and procedural complications) | 1 | 0
severe diarrhea (Gastrointestinal disorders) | 0 | 2
paraesophageal hernia (Gastrointestinal disorders) | 0 | 1
benign brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
knee replacement (Surgical and medical procedures) | 1 | 1
laminectomy (Surgical and medical procedures) | 1 | 1
repair of esophageal tear (Surgical and medical procedures) | 0 | 1
fall requiring hospitalization (Injury, poisoning and procedural complications) | 5 | 3
head injury (Injury, poisoning and procedural complications) | 0 | 1
bladder surgery (Surgical and medical procedures) | 1 | 0
eye infection (Eye disorders) | 0 | 1
hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1
medication interaction (Injury, poisoning and procedural complications) | 0 | 1
kidney or bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
abdominal pain intractable (Gastrointestinal disorders) | 1 | 0
melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
new onset overt diabetes (Endocrine disorders) | 0 | 1
detached retina (Eye disorders) | 0 | 1
cardioversion (Surgical and medical procedures) | 1 | 0
trauma (Injury, poisoning and procedural complications) | 1 | 1
gastrointestinal infection (Infections and infestations) | 0 | 2
ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
hypotension (Cardiac disorders) | 0 | 1
pacemaker placement (Surgical and medical procedures) | 1 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | Metformin (N=77)
fall (Musculoskeletal and connective tissue disorders) | 13 | 18
elevated glucose (Endocrine disorders) | 7 | 6
nausea (Gastrointestinal disorders) | 1 | 7
diarrhea (Gastrointestinal disorders) | 2 | 26
fatigue (Nervous system disorders) | 4 | 8
decreased memory (Nervous system disorders) | 0 | 4
weight loss (General disorders) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT01804049/Prot_SAP_000.pdf